CLINICAL TRIAL: NCT05767216
Title: Genetic and Epigenetic Variations in Heterokaryotypic Monozygotic Twins Discordant for Down Syndrome
Acronym: Colibri
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Jerome Lejeune (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Colibri
Record Dates: First submitted 2023-02-07; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Down syndrome children (Other): Two pairs of twins discordant for Down syndrome and 1 children with mosaic Down syndrome will be recruited. Blood, skin and feces samples will be specifically collected for the purpose of the study.
  Interventions: Other: Biological sampling

INTERVENTIONS:
Other: Biological sampling — Blood, skin and stool samples for laboratory analysis

SUMMARY:
Heterokaryotypic monozygotic twins discordant for Down syndrome (DS) are very rare, with an incidence estimated to be less than 1 over 7,000,000 pregnancy in the general population. Sharing the same genetic patrimony, except for an additional chromosome 21 for one of them, any gene-expression difference between them could be attributed only to the supernumerary chromosome 21 and not to polymorphic variability in the rest of the genome. The setting up of a prospective longitudinal study will offer the major advantage of allowing genetic and epigenetic comparisons between them and to obtain important information on the impact of the environment in which they live and grow up.

DETAILED DESCRIPTION:
It is planned to perform multi-omics analyses in order to reach an integrated understanding of the effect of genomic changes on protein expression, on biochemical posttranslational modifications of the synthetized proteins and on the modulation of some signalling pathways.

This study will also allow the generation of induced Pluripotent Stem Cells (iPSCs) from blood cells and fibroblasts of the monozygotic twins useful as in-vitro models to study the pathogenesis and the pathophysiology of Down syndrome. All this may shed the light on new research approaches in Down syndrome.

At last, the human gut microbiome, referring to the total microbial population in the human gastrointestinal tract, although thought to have its own impact, will also be studied. The microbiome is known to play a crucial role mainly in protecting the host against pathogenic microbes, modulating immunity, regulating metabolic processes, and controlling neuropsychiatric behaviour

ELIGIBILITY:
Inclusion Criteria:

* Twins of a heterokaryotypic monozygotic pair discordant for DS
* Twins of a sex- and class of age-matched dizygotic pair discordant for DS,
* Sex- and class of age-matched patient with mosaic T21
* Subject's parents/legal representatives willing to give written informed consent.
* Subject and his/her parents/legal representatives must be able/willing to comply with the protocol.
* Subject covered by social welfare.

Exclusion Criteria:

* None

Ages: 4 Years to 11 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Analysis of the coding and non-coding genetic variations between participants | 1 year
  Whole Genome Sequencing of DNA samples
Study of epigenetic modifications | 1 year
  DNA methylation pattern
Identification of active genes | 1 year
  Analysis of transcriptomic profile from RNA samples
Determination of the mechanisms of genes regulation | 1 year
  Analysis of transcriptomic profile from RNA samples
Definition of the network of genes expression | 1 year
  Analysis of transcriptomic profile from RNA samples
Identification of the proteins regulated differently | 1 year
  Analysis of proteomic profile from plasma samples
Link specific proteins to some specific complications seen in patients with Down syndrome | 1 year
  Analysis of proteomic profile from plasma samples

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jérôme Lejeune, Paris, France

IPD SHARING:
Plan to Share IPD: No